CLINICAL TRIAL: NCT01076803
Title: Prospective Study to Assess the Efficacy and Safety of Lanreotide 120 mg as a Palliative Treatment of Clinical Symptoms Associated With Malignant Intestinal Obstruction in Inoperable Patients
Brief Title: Efficacy and Safety of Lanreotide 120 Milligram (mg) as a Palliative Treatment of Clinical Symptoms Associated With Malignant Intestinal Obstruction in Inoperable Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009/289
Record Dates: First submitted 2009-12-02; First posted 2010-02-26 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Malignant Intestinal Obstruction
Keywords: Malignant intestinal obstruction in inoperable patients
MeSH Terms: interventions — lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lanreotide (acetate) (Experimental)
  Interventions: Drug: Lanreotide (acetate)

INTERVENTIONS:
Drug: Lanreotide (acetate) — Deep subcutaneous injection into the upper external quadrant of the right or the left buttock.

SUMMARY:
The primary objective of this study is to assess the efficacy of Lanreotide 120 mg for the relief of clinical symptoms due to malignant bowel obstruction in inoperable patients. This effect will be evaluated by the percentage of responder patients 7 and 14 days after one administration of lanreotide 120 mg.

(A responder patient will be defined either as a patient experiencing < or= 1 vomiting episode per day during at least three consecutive days or as a patient in whom NGT has been removed without any vomiting recurrence during at least three consecutive days)

The total number of visits will depend on the clinical situation, 5 visits are obligatory: Day(D)-3/-0,Day 1,Day 7,Day 14,Day 28

Inclusion visit (D-3/-0): eligibility, PIC, obstruction history, clinical exam, vital signs, diary cards, VAS scale, cc medication, blood sample

Visit D1: injection Visit D7/D14/28: clinical exam, nutrition procedure, result of biochemical analyse, adverse events, cc medication

In between the visits, the patient will keep and fill out his diary and VAS scale

ELIGIBILITY:
Inclusion Criteria:

* PIC
* >= 18 years at time of enrolment
* Diagnosis of a digestive obstruction of malignant origin
* Diagnosis of peritoneal carcinomatosis confirmed by a ct scan within the previous 3 months
* Inoperability as decided after surgical consultation

Exclusion Criteria:

* Operable obstruction
* Bowel obstruction that can be explained by a non malignant cause
* Signs of bowel obstruction
* Prior treatment with somatostatin analogues within the previous 60 days
* Known hypersensitivity to any of the test materials or related compounds
* Previous enrolment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Percentage of responder patients. | At day 7 and day 14.

SECONDARY OUTCOMES:
Number of daily vomiting episodes on diary cards or measurements of the daily drainage by naso gastric tube (NGT). | day 7, day 14 and day 28 after administration of Lanreotide
Number of days without vomiting episodes | day 7, day 14 and day 28 after administration of Lanreotide
Number of daily nausea episodes recorded on diary cards. | day 7, day 14 and day 28 after administration of Lanreotide
Intensity of abdominal pain assessed on a visual analogue scale. | day 7, day 14 and day 28 after administration of Lanreotide.
Well-being assessed on a visual analogue scale. | day 7, day 14 and day 28 after administration of Lanreotide.
Time between first injection and clinical response. | day 7, day 14 and day 28 after administration of Lanreotide
Clinical and biological adverse events. | day 7, day 14 and day 28 after administration of Lanreotide.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Geboes, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website of the University Hospital Ghent — http://www.uzgent.be